CLINICAL TRIAL: NCT04064125
Title: A 21-Day, Randomized, Controlled Study to Evaluate the Skin Irritation Potential of FMX-101 in Healthy Volunteers Using a Cumulative Irritant Patch Test Design
Brief Title: Dermal Cumulative Irritant Patch Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX2016-08
Record Dates: First submitted 2019-08-08; First posted 2019-08-21 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Healthy
MeSH Terms: interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FMX-101 (Experimental)
  Interventions: Drug: FMX-101

INTERVENTIONS:
Drug: FMX-101

SUMMARY:
A 21-Day, Randomized, Controlled Study to Evaluate the Skin Irritation Potential of FMX-101 in Healthy Volunteers Using a Cumulative Irritant Patch Test Design

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females who were 18 years of age or older.
* Were of any Fitzpatrick Skin Type or race, providing the skin pigmentation allowed for discernment of erythema.

Exclusion Criteria:

* Had any visible skin disease at the application site which, in the opinion of the investigative personnel, would have interfered with the evaluation of the test site reaction.
* Had damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-10-28 (Actual)

PRIMARY OUTCOMES:
Comparison of mean cumulative irritation over time for IP versus controls using a dermal irritation numerical equivalent grading tool. | 3 weeks